CLINICAL TRIAL: NCT02712333
Title: Health Effects of Indoor Air Filtration in Healthy Chinese Adults: An Intervention Study
Brief Title: Health Effects of Indoor Air Filtration in Healthy Chinese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FDEH-AF2015
Record Dates: First submitted 2016-02-01; First posted 2016-03-18 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-05

CONDITIONS: Blood Pressure
Keywords: PM2.5; air purification; randomized controlled trial; metabolomics; Metabolites; exhaled nitric oxide
MeSH Terms: interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Air purifiers (Experimental): Participants in this group received an intervention of true air purifiers placed in the center of the room.
  Interventions: Behavioral: Air Purifiers
- Control (Sham Comparator): Participants in this group received an intervention of sham air purifiers, which were under the same conditions as the true purifiers except the filter gauze in them were removed.
  Interventions: Behavioral: Sham Air Purifiers

INTERVENTIONS:
Behavioral: Air Purifiers — The 17 dormitory rooms and their residents were randomized into two groups: the intervention and control group. The intervention group went through a 9-day intervention with an air purifier placed in the center of the room. All rooms in this group used the same qualified air purifiers (model KJEA200e, 3M), and all participants were required to stay in their dormitory rooms with the windows/doors closed throughout intervention period. All participants and research staffs were blinded to the group assignment.
  Arms: Air purifiers
Behavioral: Sham Air Purifiers — The control group went through a 9-day intervention with a sham air purifier (with its filter gauze removed) placed in the center of the room. All rooms used the same air purifiers (model KJEA200e, 3M) as the intervention group, except the filter gauze was removed. During the study period all participants were required to stay in their dormitory rooms with the windows/doors closed. All participants and research staffs were blinded to the group assignment.
  Arms: Control

SUMMARY:
This study aims to detect serum metabolite changes, as well as other health indicators with the intervention of air purifiers on a randomized, crossover, double-blind trial.

DETAILED DESCRIPTION:
The investigators conducted a randomized double-blind crossover trial among 60 healthy college students in Shanghai, China from November to December, 2015. These students lived in dormitories that were randomized into two groups and alternated the use of true or sham air purifiers for 9 consecutive days with a 2-week wash-out interval. All participants and research staffs were blinded to the group assignment. All participants were required to stay in their dormitory with the windows/doors closed for at least 50% of the time on weekdays and for 80% on weekends throughout the 9-day intervention period. All interventions started at 7 a.m. to avoid issues related to diurnal variation. Health endpoints, including blood pressure, fractional exhaled nitric oxide were evaluated and biological samples such as morning urine, fast blood and buccal cells were collected at baseline and immediately after the completion of each intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy university students in Jiangwan Campus, Fudan university
* Non-smoking, no history of alcohol or drug abuse
* Free of chronic cardiovascular, respiratory, liver and kidney disease
* Spend at least 50% (weekdays) or 80% (weekends) of time indoors

Exclusion Criteria:

* Current or ever smokers
* History of asthma, chronic bronchitis，cough, hypertension or other chronic inflammatory disease
* acute infections
* medication use in recent one month

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, Ph.D., Study Director — School of Public Health，Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li H, Cai J, Chen R, Zhao Z, Ying Z, Wang L, Chen J, Hao K, Kinney PL, Chen H, Kan H. Particulate Matter Exposure and Stress Hormone Levels: A Randomized, Double-Blind, Crossover Trial of Air Purification. Circulation. 2017 Aug 15;136(7):618-627. doi: 10.1161/CIRCULATIONAHA.116.026796. PMID 28808144

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted on November, 2015 in Jiangwan Campus, Fudan University. A total of 65 participants were assessed for eligibility and 60 of them were finally recruited
Groups:
- Group 1-air Purification First, Then Sham Air Purification: Participants in this group received an intervention of true air purifiers placed in the center of the room.
  Real Air Purification: The 17 dormitory rooms and their residents were randomized into two groups: the intervention and control group. The intervention group went through a 9-day intervention with an air purifier placed in the center of the room. All rooms in this group used the same qualified air purifiers (model KJEA200e, 3M), and all participants were required to stay in their dormitory rooms as much as possible with the windows/doors closed throughout intervention period. All participants and research staffs were blinded to the group assignment.
- Group2-sham Air Purification First, Then Real Air Purification: Participants in this group received an intervention of sham air purifiers, which were under the same conditions as the true purifiers except the filter gauze in them were removed.
  Sham Air Purification: This group went through a 9-day intervention with a sham air purifier (with its filter gauze removed) placed in the center of the room. All rooms used the same air purifiers (model KJEA200e, 3M) as the intervention group, except the filter gauze was removed. During the study period all participants were required to stay in their dormitory rooms as much as possible with the windows/doors closed. All participants and research staffs were blinded to the group assignment.
Period: First Period
Arm/Group | Group 1-air Purification First, Then Sham Air Purification | Group2-sham Air Purification First, Then Real Air Purification
Started | 34 | 26
Completed | 31 | 24
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2
Period: Second Period
Arm/Group | Group 1-air Purification First, Then Sham Air Purification | Group2-sham Air Purification First, Then Real Air Purification
Started | 31 | 24
Completed | 31 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group1-air Purification First, Then Sham Air Purification: Participants in this group received a treatment of true air purification first, and then switched to the sham purification treatment the second stage.
  For real air purification, we used high efficient air purifiers (model KJEA200e, 3M), and all participants were required to stay in their dormitory rooms with the windows/doors closed throughout intervention period. For sham air purification, we placed a sham air purifier (with HEPA filters removed) while keeping the rest of the experiment conditions and requirements for the participants unchanged. All participants and research staffs were blinded to the group assignment.
- Group2-sham Air Purification First, Then Real Air Purification: Participants in this group received a treatment of sham air purification first, and then switched to the real purification treatment the second stage.
  For real air purification, we used high efficient air purifiers (model KJEA200e, 3M), and all participants were required to stay in their dormitory rooms with the windows/doors closed throughout intervention period. For sham air purification, we placed a sham air purifier (with HEPA filters removed) while keeping the rest of the experiment conditions and requirements for the participants unchanged. All participants and research staffs were blinded to the group assignment.
- Total: Total of all reporting groups
Arm/Group | Group1-air Purification First, Then Sham Air Purification | Group2-sham Air Purification First, Then Real Air Purification | Total
Number analyzed (Participants) | 31 | 24 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.0 (1.3) | 20.6 (1.4) | 20.2 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 14 | 13 | 27
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 21.6 (2.9) | 20.6 (2.5) | 21.1 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Changes of Serum Cortisol Levels
Description: Using metabolomic methods to screen and quantify all the serum metabolites, and calculate changes in main metabolites in sham purification compared to real purification.
  Relative intensity was calculated by dividing the peak intensity of cortisol with the peak intensity of internal standard (2-chloro-D-phenylalanine methanol solution, 0.014mg/mL)
Time Frame: at the end of each 9-day intervention period
Measure: Mean (Standard Deviation); unit: relative intensity
Groups:
- Real Purification: Participants in this group received a treatment of air purification.
- Sham Purification: Participants received sham air purification first.
Arm/Group | Real Purification | Sham Purification
Number analyzed (Participants) | 55 | 55
relative intensity | 0.012835 (0.00371) | 0.016206 (0.00474)
Statistical Analysis 1: Comparison: Real Purification vs Sham Purification; we analyzed the serum cortisol levels (presented as relative intensities in high perfomance liquid chromatography-mass spectrum) by treatments (intervention group vs control group); Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — the p-value has been adjusted for multiple comparisons; % increase per 10μg/m3 increase of PM2.5 = 7.53, 95% CI 2-sided [4.65 to 10.41]
Statistical Analysis 2: Comparison: Real Purification vs Sham Purification; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; fold change = 1.33 — fold change is calculated by measurments from the sham purification group/measurements from the real purification group

2. Primary Outcome: Changes of Serum Cortisone Concentration
Description: Use metabolomic methods to screen and quantify all the serum metabolites, and calculate changes in main metabolites in sham purification compared to real purification.
  Relative intensity was calculated by dividing the peak intensity of cortisone with the peak intensity of internal standard (2-chloro-D-phenylalanine methanol solution, 0.014mg/mL)
Time Frame: at the end of each 9-day intervention period
Measure: Mean (Standard Error); unit: relative intensity
Groups:
- Real Purification: Participants received a treatment of air purification
- Sham Purification: Participants received a treatment of sham air purification
Arm/Group | Real Purification | Sham Purification
Number analyzed (Participants) | 55 | 55
relative intensity | 0.021076 (0.004375) | 0.024338 (0.004625)
Statistical Analysis 1: Comparison: Real Purification vs Sham Purification; we analyzed the serum cortisone levels by treatment (intervention group vs control group); Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — the p-value has been adjusted for multiple comparisons; % increase per 10μg/m3 increase of PM2.5 = 3.69, 95% CI 2-sided [1.85 to 5.54]
Statistical Analysis 2: Comparison: Real Purification vs Sham Purification; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; fold change = 1.18 — fold change is calculated by measurments from the sham purification group/measurements from the real purification group

3. Primary Outcome: Changes of Serum Epinephrine Concentrations
Description: Use metabolomic methods to screen and quantify all the serum metabolites, and calculate changes in main metabolites in sham purification compared to real purification.
  Relative intensity was calculated by dividing the peak intensity of epinephrine with the peak intensity of internal standard (2-chloro-D-phenylalanine methanol solution, 0.014mg/mL)
Time Frame: at the end of each 9-day intervention
Measure: Mean (Standard Error); unit: relative intensity
Groups:
- Real Purification: Participants received a treatment of real air purification.
- Sham Air Purification: Participants received a treatment of sham air purification.
Arm/Group | Real Purification | Sham Air Purification
Number analyzed (Participants) | 55 | 55
relative intensity | 0.140609 (0.027514) | 0.165321 (0.036633)
Statistical Analysis 1: Comparison: Real Purification vs Sham Air Purification; we analyzed the serum epinephrine levels by treatment (intervention group vs control group); Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — the p-value has been adjusted for multiple comparisons; % increase per 10μg/m3 increase of PM2.5 = 5.17, 95% CI 2-sided [3.21 to 7.14]
Statistical Analysis 2: Comparison: Real Purification vs Sham Air Purification; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; fold change = 1.20 — fold change is calculated by measurments from the sham purification group/measurements from the real purification group

4. Primary Outcome: Changes of Serum Norepinephrine Concentration
Description: Use metabolomic methods to screen and quantify all the serum metabolites, and calculate changes in main metabolites in sham purification compared to real purification.
  Relative intensity was calculated by dividing the peak intensity of cortisol with the peak intensity of internal standard (2-chloro-D-phenylalanine methanol solution, 0.014mg/mL)
Time Frame: at the end of each 9-day intervention
Measure: Mean (Standard Deviation); unit: relative intensity
Arm/Group | Real Purification | Sham Purification
Number analyzed (Participants) | 55 | 55
relative intensity | 0.030752 (0.024335) | 0.038695 (0.024624)
Statistical Analysis 1: Comparison: Real Purification vs Sham Purification; we analyzed the serum norepinephrine levels by treatment (intervention group vs control group); Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — the p-value has been adjusted for multiple comparisons; % increase per 10μg/m3 increase of PM2.5 = 11.28, 95% CI 2-sided [7.37 to 15.21]
Statistical Analysis 2: Comparison: Real Purification vs Sham Purification; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; fold change = 1.57 — fold change is calculated by measurments from the sham purification group/measurements from the real purification group

5. Secondary Outcome: Systolic Blood Pressure
Description: To eliminate possible error, blood pressure for each participant were conducted by the same working staff using the same instrument. Average levels were calculated by treatments (intervention or control).
Time Frame: at the end of each 9-day intervention period
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Real Purification | Sham Purification
Number analyzed (Participants) | 55 | 55
mmHg | 102.2 (13.4) | 104.8 (12.8)
Statistical Analysis 1: Comparison: Real Purification vs Sham Purification; we analyzed the serum SBP levels by treatment (intervention group vs control group); Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; % increase per 10μg/m3 increase of PM2.5 = 0.84, 95% CI 2-sided [0.09 to 1.59]

6. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 5
Time Frame: at the end of each 9-day intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Real Purification | Sham Air Purification
Number analyzed (Participants) | 55 | 55
mmHg | 64.5 (9.6) | 65.2 (8.8)
Statistical Analysis 1: Comparison: Real Purification vs Sham Air Purification; we analyzed the serum cortisol levels by treatment (intervention group vs control group); Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; % increase per 10μg/m3 increase of PM2.5 = 0.31, 95% CI 2-sided [-1.59 to 0.96]

7. Secondary Outcome: Pulse Pressure
Description: as for outcome 5
Time Frame: at the end of each 9-day intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Real Purification | Sham Air Purification
Number analyzed (Participants) | 55 | 55
mmHg | 37.7 (7.5) | 39.6 (8.3)
Statistical Analysis 1: Comparison: Real Purification vs Sham Air Purification; we analyzed the serum cortisol levels by treatment (intervention group vs control group); Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; % increase per 10μg/m3 increase of PM2.5 = 1.24, 95% CI 2-sided [-1.14 to 3.63]

ADVERSE EVENTS:
Groups:
- Real Air Purification: Participants in this group received an intervention of true air purifiers placed in the center of the room.
  Real Air Purification: The 17 dormitory rooms and their residents were randomized into two groups: the intervention and control group. The intervention group went through a 9-day intervention with an air purifier placed in the center of the room. All rooms in this group used the same qualified air purifiers (model KJEA200e, 3M), and all participants were required to stay in their dormitory rooms as much as possible with the windows/doors closed throughout intervention period. All participants and research staffs were blinded to the group assignment.
- Sham Air Purification: Participants in this group received an intervention of sham air purifiers, which were under the same conditions as the true purifiers except the filter gauze in them were removed.
  Sham Air Purification: This group went through a 9-day intervention with a sham air purifier (with its filter gauze removed) placed in the center of the room. All rooms used the same air purifiers (model KJEA200e, 3M) as the intervention group, except the filter gauze was removed. During the study period all participants were required to stay in their dormitory rooms as much as possible with the windows/doors closed. All participants and research staffs were blinded to the group assignment.
Arm/Group | Real Air Purification | Sham Air Purification
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No